CLINICAL TRIAL: NCT06353789
Title: Understanding the Role of Adolescent Dysmenorrhoea as a Risk Factor for the Transition to Chronic Pain: Clinical Cohort Study
Brief Title: Adolescent Dysmenorrhoea as a Risk Factor for Chronic Pain: Clinical Cohort Study
Acronym: RoADPain
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Exeter (Other); University of York (Other); Endometriosis UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: RoADPain Clinical Study
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-04

CONDITIONS: Dysmenorrhea
Keywords: Adolescent; chronic pain
MeSH Terms: conditions — Dysmenorrhea; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva will be collected and genotyping undertaken
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysmenorrhoea: Reports period pain ≥4/10 and no other chronic pain
- Controls: Reports period pain ≤3/10 and no other chronic pain

SUMMARY:
This study aims to understand whether changes in a variety of body systems which are seen in adult women with period pain are also seen in adolescents in the first few years of having periods. This information will help to understand 1) how quickly any changes occur, informing clinical practice, and 2) how period pain might lead to other types of chronic pain, potentially allowing development of preventative strategies.

DETAILED DESCRIPTION:
Chronic pain is defined as pain that lasts for more than 3 months. It is really common, affecting up to 30% of people worldwide with impacts on all areas of life. Chronic pain is difficult to treat once it has developed. Therefore, understanding which people might be at risk of developing chronic pain and protecting them from it starting, would be a really positive step forward.

It is known that women are more likely to develop almost all types of chronic pain than men. This sex difference in chronic pain starts to be seen after puberty, suggesting that changes happening at this time may be contributing to this increased risk. One important change that happens at this time is periods starting. Despite periods often being very painful, period pain has traditionally been dismissed as "normal" and something girls must learn to live with. However, in adult women with period pain many differences are seen across a range of body systems when compared to women without period pain. These include increased sensitivity to pain; increased sensitivity of the bladder, bowel and womb; altered brain structure and function; and altered responses to stress. Similar changes to those seen with period pain can be seen in other chronic pain conditions. It is not known whether these changes are caused by repeated or continuous pain or if they are part of the reason why chronic pain develops, or a combination of both.

The RoADPain Clinical Study aims to see whether the differences in other body systems described above in adult women with period pain are also seen in girls in the first few years of having periods. The investigators will combine detailed questionnaire data with tests of the function of a variety of systems (including nerve function, stress response and brain imaging). No study treatment or intervention will be given. It is envisaged that this information will help to understand 1) how quickly any changes occur, informing clinical practice, and 2) how period pain might lead to other types of chronic pain, potentially allowing development of preventative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or parent/guardian of participant) is willing and able to give informed consent for participation in the study.
* Female or assigned female at birth.
* aged 11 - 20 years.
* At least 6 periods per year since menarche.
* During the study data collection period will be within one of the following time intervals since menarche:
* 12 - 15 months
* 36 - 39 months
* 60 - 63 months
* Reports either period pain or no pain with periods and scores appropriately on NRS (period pain: ≥4/10; no period pain: ≤3/10).
* Not using hormonal therapies (i.e. contraceptives) currently and has not used previously.
* Reasonably fluent in English.

Exclusion Criteria:

* Current or previous chronic pain condition other than dysmenorrhoea, including migraine.
* Pregnant or breast-feeding.
* Previous cancer diagnosis.
* Contraindication to MRI

Ages: 11 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Sensory Testing (QST) | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  QST of the left hand according to the German Neuropathic Pain Network Protocol plus an auditory stimulus.
Heart rate (HR) | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Assessed over a 20 minute period at rest.
Change in heart rate | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Assessed at rest immediately before the CPM paradigm described below and then again immediately after. The ischaemic pain stimulus used as the conditioning stimulus in this paradigm is the most noxious component of the physiological testing paradigms used in this study and therefore the most likely to generate a stress response. The change will be reported as HR(before) - HR(after).
Bladder sensitivity to filling | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Assessed with standardised non-invasive bladder filling paradigm, measured as time to verbal reports of different sensations of bladder fullness (first sensation, first urge) and then need to void (maximum tolerance) after drinking 600 ml water. Subjects will be categorised into those with bladder sensitivity compared to published norms for similar age adolescents and those with normal bladder sensation.
Volume voided at maximum tolerance | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Assessed with standardised non-invasive bladder filling paradigm described in outcome 4. The volume of urine voided when maximum tolerance is reached will be measured in mls.
Pain Catastrophising: Pain Catastrophising Scale (PCS) (Sullivan) | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Measured with the Pain Catastrophising Scale (Sullivan). Scores range from 0 - 52 with high scores representing higher levels of pain catastrophising. Although three sub scales exist they will not be assessed for the purposes of these main analyses.
Area under the curve (AUC) of single day salivary cortisol profile | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  Saliva will be collected at home at the specified times allowing a daily AUC of salivary cortisol for each subject to be calculated. Collection times: waking; 30-45 minutes after waking; before lunch; before dinner; bedtime.

SECONDARY OUTCOMES:
Change of pressure pain threshold (PPT) | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  A standardised conditioned pain modulation (CPM) paradigm will be used to investigate the change in pressure pain threshold on the dorsum of the foot. An ischaemic stimulus to the contralateral arm will be used as the conditioned stimulus. The foot PPT will be measured before the conditioned stimulus and immediately after. The change will be reported as the (PPTbefore - PPTafter).
fMRI scan | days 1-3 (menstrual phase) and days 10-12 (follicular phase) of the menstrual cycle.
  fMRI scan with resting sequences, response to punctate stimulation of the abdomen and visual stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Katy Vincent, MRCOG, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the study and all follow up analyses are complete de-identified data will be deposited in a publically accessible repository as required by the funders.
Supporting Information: Study Protocol
Time Frame: Data will be available once all analyses are complete.
Access Criteria: Data will be publically accessible